CLINICAL TRIAL: NCT05862714
Title: Comparison of Efficacy of Single Oral Dose Fluconazole and Itraconazole in Patients With Pityriasis Versicolor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr Aleena Nasir, Principal Investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMHAbbottabad1
Record Dates: First submitted 2023-03-30; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Tinea Versicolor
MeSH Terms: conditions — Tinea Versicolor | interventions — Fluconazole; Itraconazole; icon infiltrant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Fluconazole (Active Comparator): Oral fluconazole (400 mg stat) given to patients.
  Interventions: Drug: Fluconazole; Drug: Itraconazole
- Group B Itraconazole (Active Comparator): Oral Itraconazole (1000 mg stat) given to patients.
  Interventions: Drug: Fluconazole; Drug: Itraconazole

INTERVENTIONS:
Drug: Fluconazole — 400 mg stat. Follow up at 4 weeks
  Other Names: Fluderm
Drug: Itraconazole — 1000 mg stat. Follow up at 4 weeks
  Other Names: Icon

SUMMARY:
Pityriasis versicolor (PV) also called tinea versicolor is a common superficial chronic fungal infection of the skin caused by species of lipophilic yeast known as Malassezia species. Itraconazole is an oral synthetic triazole while fluconazole is an oral synthetic bis-triazole compound. Only a few studies are available to find a direct comparison of the efficacy of single dose of oral fluconazole (400 mg) and oral itraconazole (1000 mg) in the treatment of PV. The objective of the study was to compare the efficacy of single dose fluconazole (400 mg stat) to single dose itraconazole (1000 mg stat) in the treatment of pityriasis versicolor in the local population of Pakistan.

DETAILED DESCRIPTION:
Pityriasis versicolor (PV) also called tinea versicolor is a common superficial chronic fungal infection of the skin caused by species of lipophilic yeast known as Malassezia species. Itraconazole is an oral synthetic triazole while fluconazole is an oral synthetic bis-triazole compound. These both acts by inhibiting the cytochrome-P450 dependent 14-alpha-demethylation step in the formation of ergosterol thereby impairing the functions of certain membrane bound enzyme systems, and ultimately inhibiting the growth of fungi. Both the drugs have been studied in different dose regimen, however, there are variable results in studies on this subject. There is still no standard drug and its dosage that can ensure complete cure. Fluconazole (300mg) in 2 doses with an interval of one week has been used effectively, however, fluconazole (400 mg) as a single dose has also been used, and found to cure the PV. Itraconazole 200 mg/day can be given in a dose of for 7 days however, higher concentrations of itraconazole in the stratum corneum are achieved that persist for 3-4 weeks so the drug is presumed to be effective even in a single dose. Therefore, only a few studies are available to find a direct comparison of the efficacy of single dose of oral fluconazole (400 mg) and oral itraconazole (1000 mg) in the treatment of PV. The objective of the study was to compare the efficacy of single dose fluconazole (400 mg stat) to single dose itraconazole (1000 mg stat) in the treatment of pityriasis versicolor in the local population of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* All the patients above 18 years of age
* Diagnosed with pityriasis versicolor

Exclusion Criteria:

* Those patients who had received any antifungal treatment during last 1 month
* pregnancy
* lactation
* history of renal disease hepatic disease or malignancy
* history of hepatic disease
* history of malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement Resolution of symptoms | 4 weeks
  Efficacy of treatment was assessed by mycological test by making KOH mount at start of treatment and than at follow up at 4 weeks
Efficacy of treatment through KOH mount | 4 weeks
  Efficacy of treatment was assessed by mycological test by making KOH mount at start of treatment and than at follow up at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Abbottabad, Abbottābād, Khyber Pakhtunkhwa, Pakistan